CLINICAL TRIAL: NCT00163566
Title: A Phase II, Placebo-Controlled, Double-Blind, Dose-Ranging (35mg/Day or 70 mg/Day), Randomized, Study of Cutaneous Dihydrotestosterone (DHT)-Gel (0.7% Hydroalcoholic Gel) in Older Hypogonadal Males Ages 55-80 Years: Effect on Body Composition, Libido, and Physical and Sexual Functioning
Brief Title: Study of DHT-Gel to Treat the Symptoms of Low Testosterone in Men 55-80
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASCEND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-DHT-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Hypogonadism; Late Onset Hypogonadism; Low Testosterone
Keywords: libido; depression strength; testosterone; dihydrotestosterone
MeSH Terms: conditions — Hypogonadism | interventions — Dihydrotestosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Placebo gel (Placebo Comparator): Placebo gel twice per day
  Interventions: Drug: Dihydrotestosterone (0.7%) in hydroalcoholic gel
- 0.7% DHT gel, Dose 1 (Active Comparator): 0.7% DHT gel twice per day, 35 mg/day
  Interventions: Drug: Dihydrotestosterone (0.7%) in hydroalcoholic gel
- 0.7% DHT gel, Dose 2 (Active Comparator): 0.7% DHT gel twice per day, 70 mg/day
  Interventions: Drug: Dihydrotestosterone (0.7%) in hydroalcoholic gel

INTERVENTIONS:
Drug: Dihydrotestosterone (0.7%) in hydroalcoholic gel — transdermal gel, 0.7% DHT, 0.35 mg/day or 0.70 mg/day total daily dose (or placebo gel), applied twice per day

SUMMARY:
The purpose of this study is to evaluate whether DHT-Gel, when applied daily to the skin, can relieve the symptoms of low testosterone in men aged 55-80. These symptoms include reduced muscle strength, increase fat mass, low libido, feeling blue or moody

DETAILED DESCRIPTION:
Background - In the context of hypogonadism, androgen supplementation is clearly beneficial, particularly in younger males. The benefits of therapy in men with milder degrees of hypogonadism, and elderly males with testosterone deficiency, are less clear-cut. Several options are available for androgen replacement in adult men. Oral testosterone, intramuscular injections, subcutaneous implants and transdermal therapy have all been used. Each mode of delivery has advantages and drawbacks. Several alkylated derivatives of T are available for oral or sublingual use, including methyl testosterone and fluoxymesterone. However, they are not recommended for use as replacement therapy because of their associated adverse effects.

Study Design - This is a multi-center, double-blind, placebo-controlled, parallel group, randomized study of DHT-Gel versus placebo gel in male subjects ages 55-80 years inclusive with low serum testosterone and symptoms compatible with the clinical diagnosis of hypogonadism. Total enrollment for this study will be approximately 120 subjects (40 subjects for each treatment group). Subjects will be treated with 35 mg/day DHT, 70 mg/day DHT, or placebo gel for 6 months. All subjects will apply the gel once daily. Up to 9 months of study participation, including up to 2 months of screening and a 1-month follow-up period, will be required by the protocol.

The primary efficacy endpoint in this study is change in body composition as determined by DEXA scan. Secondary endpoints in this study include change in sexual libido, and overall function and mood, and normalization of serum androgen levels. A subset of sites will perform strength assessments, which will include handgrip dynamometry, and upper and lower body strength tests.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 55-80 Serum Testosterone < 275 Symptoms of Hypogonadism as determined by AMS scale In good overall health

Exclusion Criteria:

* Abnormal Prostate Exam for age Prostate or Breast Cancer Significant illness Weight >300lbs Generalized skin disease Unstable sleep apnea

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2004-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Body Composition

SECONDARY OUTCOMES:
Change in sexual libido, and overall function and mood
Normalization of serum androgen levels

CONTACTS AND LOCATIONS:
Overall Officials: Neta R Nelson, Study Director — ASCEND Therapeutics
Locations (16):
- United States (16):
  - Radiant Research - Phoenix, Phoenix, Arizona
  - Harbor UCLA Medical Reserach and Education Institute, Torrance, California
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Genesis Research Consultants, Longwood, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - North Indiana Research, Fort Wayne, Indiana
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Bethesda Health Research, Bethesda, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health Sciences Center, Portland, Oregon
  - VA Medical Center, Houston, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - McGuire VA Medical Center, Richmond, Virginia
  - VA Puget Sound Health Care, Seattle, Washington